CLINICAL TRIAL: NCT04227743
Title: Evaluation of Safety and Diagnostic Yield of Cryobiopsy Versus Forceps Biopsy in Endobronchial Lesions:Assiut University Experience
Brief Title: Safety and Diagnostic Yield of Cryobiopsy Versus Forceps Biopsy in Endobronchial Lesions:Assiut University Experience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Sayed Khalifa, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cryobiopsy
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-01

CONDITIONS: Endobronchial Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with endobronchial lesions (Experimental): flexible bronchoscoy will be performed to patients with endobronchial lesions and biopsy from the lesions by forceps and cryoprope will be obtained
  Interventions: Device: cryobiopsy

INTERVENTIONS:
Device: cryobiopsy — . The cryobiopsy samples will be obtained by advancement of the cryoprobe into the working channel of the bronchoscope to touch the tip of the endobronchial tumor. The freezing time will be approximately 4 seconds. Then, flexible bronchoscope together with tissue sample attached to the tip of the frozen probe will be extracted outside the bronchial tree. The tissue sample will be released from the probe's tip by plunging it into saline at room temperature. FB will be reintroduced after cryobiopsy to evaluate and control the bleeding.

SUMMARY:
The purpose of this study is to assess the diagnostic yield and show the feasibility and safety of endobronchial biopsies using the flexible cryoprob and to assess the sensitivity of cryobiopsy compared with forceps biopsy

DETAILED DESCRIPTION:
Flexible bronchoscopy is the diagnostic tool of choice to diagnose endobronchial malignancies. It allows inspection and biopsy of any endobronchial abnormalities under direct vision.

One of the main goals of diagnostic bronchoscopy, besides visualization of endobronchial abnormalities, is obtaining an adequate tissue samples from the suspicious lesions for cytohistological examination. Several techniques could be applied through the working channel of the ﬂexible bronchoscopy such as forceps biopsy, brush, bronchial washing and transbronchial needle aspiration.Flexible bronchoscopy and the associated tissue sampling techniques are the most widespread procedures in the diagnosis of central lung cancer. Even though the specimens are obtained under direct vision, there is a significant failure rate, which therefore, requires repeated bronchoscopies. Concurrent application of different sampling techniques at bronchoscopy has been shown to improve the yield.

Diagnostic bronchoscopy with endobronchial forceps biopsy is primarily practiced in patients with suspected thoracic malignancy and visible endobronchial.

The major drawback of the forceps biopsy technique is the relatively small amount of tissue obtained, which is determined by the size of the forceps. Additionally, mechanical compression or crush artefacts from the instrument tip cause alterations of the tissue samples, which affect the quality of the histological analysis. Flexible cryoprobes were introduced as a new tool for bronchoscopic tissue sampling. It is used primarily for debulking and cryoextraction of malignant airway stenosis.

With this technique, the sample is collected while still being frozen with the tissue attached on the frozen tip of the probe. By this way, larger tissue samples can be taken from endobronchial lesions and artifact free. The molecular markers are also ions. Tissue samples obtained with cryoprobes are of good quality, size better preserved and well represented.

ELIGIBILITY:
Inclusion Criteria:

- 1. Exophytic endobronchial tumor (endoscopically visible lesion)

3.Age>18 years old

Exclusion Criteria:

- 1.Patients, who refused to be included in this study or unfit for flexible bronchoscopy 2.patients with hemorrhagic diathesis (prothrombin concentration <50% and platelet count <80,000/mm 3).

3.Suspected connection of the lesion to large pulmonary blood vessels as seen on chest computed tomography scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
. Assess the diagnostic yield and show the feasibility and safety of endobronchial biopsies using the flexible cryoprobe. | 1 year
  size (im millimeter) of biopsy from endobronchial lesion obtained by cryoprobe in comparison to those obtained bu flexible forceps

SECONDARY OUTCOMES:
complication assessment | 1 year
  Post interventional bleeding classifed into:
  * No bleeding -Mild bleeding, which was controlled by maintained suction.-
  * Moderate bleeding, which can be controlled with different interventional techniques e.g local application of saline either normal or cold, adrenalin or balloon tamponade
  * Severe bleeding, which necessitates ICU admission due to hemodynamic instability and required blood transfusion

REFERENCES:
- [Background] Dobler CC, Crawford AB. Bronchoscopic diagnosis of endoscopically visible lung malignancies: should cytological examinations be carried out routinely? Intern Med J. 2009 Dec;39(12):806-11. doi: 10.1111/j.1445-5994.2008.01882.x. PMID 20233241
- [Background] Rivera MP, Detterbeck F, Mehta AC; American College of Chest Physicians. Diagnosis of lung cancer: the guidelines. Chest. 2003 Jan;123(1 Suppl):129S-136S. doi: 10.1378/chest.123.1_suppl.129s. PMID 12527572
- [Background] Schreiber G, McCrory DC. Performance characteristics of different modalities for diagnosis of suspected lung cancer: summary of published evidence. Chest. 2003 Jan;123(1 Suppl):115S-128S. doi: 10.1378/chest.123.1_suppl.115s. PMID 12527571
- [Background] Hetzel M, Hetzel J, Schumann C, Marx N, Babiak A. Cryorecanalization: a new approach for the immediate management of acute airway obstruction. J Thorac Cardiovasc Surg. 2004 May;127(5):1427-31. doi: 10.1016/j.jtcvs.2003.12.032. PMID 15116003
- [Background] Schumann C, Hetzel J, Babiak AJ, Merk T, Wibmer T, Moller P, Lepper PM, Hetzel M. Cryoprobe biopsy increases the diagnostic yield in endobronchial tumor lesions. J Thorac Cardiovasc Surg. 2010 Aug;140(2):417-21. doi: 10.1016/j.jtcvs.2009.12.028. Epub 2010 Mar 11. PMID 20226474
- [Background] Babiak A, Hetzel J, Krishna G, Fritz P, Moeller P, Balli T, Hetzel M. Transbronchial cryobiopsy: a new tool for lung biopsies. Respiration. 2009;78(2):203-8. doi: 10.1159/000203987. Epub 2009 Feb 21. PMID 19246874
- [Background] Aktas Z, Gunay E, Hoca NT, Yilmaz A, Demirag F, Gunay S, Sipit T, Kurt EB. Endobronchial cryobiopsy or forceps biopsy for lung cancer diagnosis. Ann Thorac Med. 2010 Oct;5(4):242-6. doi: 10.4103/1817-1737.69117. PMID 20981186